CLINICAL TRIAL: NCT02927990
Title: Contrast Volume Reduction During Percutaneous Coronary Interventions With the Use of a New Assisting Software Package
Brief Title: Contrast Volume Reduction During PCI With the Use of a New Assisting Software Package
Status: Terminated | Type: Observational
Why Stopped: Insights and learnings were used to initiate an improved multicenter study.
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: XCY607-130198
Record Dates: First submitted 2016-09-23; First posted 2016-10-07 (Estimated); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Coronary Stenosis; Coronary Occlusion
MeSH Terms: conditions — Coronary Stenosis; Coronary Occlusion | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group: Percutaneous coronary interventions with additional imaging provided by the new software package
  Interventions: Other: Percutaneous Coronary Intervention
- Control group: Percutaneous coronary interventions without the new software package
  Interventions: Other: Percutaneous Coronary Intervention

INTERVENTIONS:
Other: Percutaneous Coronary Intervention — Percutaneous Coronary Intervention according to standard of care

SUMMARY:
The new software package is intended to assist the physician in imaging the coronaries during percutaneous coronary interventions.

This study investigates the amount of contrast used during percutaneous coronary interventions with the aid of the new software package.

The results of the study will be compared with control group data (before the new software package was installed or after it was removed) to define a possible contrast reduction.

ELIGIBILITY:
Inclusion Criteria:

* Subject undergoing a percutaneous coronary intervention.
* Subject 18 years of age or older, or of legal age to give informed consent per state or national law.

Exclusion Criteria:

* Subject undergoing an emergency treatment
* Primary angioplasty for acute ST segment elevation myocardial infarction.
* Subject with contrast allergies
* Subject with severe kidney disease (e-GFR < 40 by Modification of Diet in Renal Disease (MDRD)/Cockcroft Gault clearance formula and/or upon decision by investigator)
* Subject participates in a potentially confounding drug or device trial during the course of the study.
* Prisoners, people who cannot legally give consent, pregnant women and breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with age 18 or older, of both genders and all races. Patients undergoing a percutaneous coronary intervention. Patients are considered to be enrolled in the study after they have signed the informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Parikh, MD, Principal Investigator — Columbia University Medical Center/NYPH
Locations (1):
- Columbia University Medical Center/NYPH, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 subjects are enrolled. Phase 2 not initiated.
Groups:
- Subject Undergoing PCI Phase 1: Subject undergoing a percutaneous coronary intervention with navigation support of Dynamic Coronary Roadmap
Period: Overall Study
Arm/Group | Subject Undergoing PCI Phase 1
Started | 80
Completed | 24
Not Completed | 56
Not completed — Protocol Violation | 4
Not completed — Physician Decision | 9
Not completed — Room switched and therefore no study device available | 15
Not completed — No procedure performed, only diagnostic catheterization | 28

BASELINE CHARACTERISTICS:
Arm/Group | Subject Undergoing PCI Phase 1
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Amount [mL] of Contrast Used for Completion of the Coronary Intervention
Description: Phase 2 not initiated Only phase 1 data was collected
Time Frame: Amount of contrast [mL] will be determined once, at the end of the Percutaneous Coronary Intervention. There is no patient follow-up.
Population: No data gathered for the primary outcome. Phase 2 not initiated Only phase 1 data was collected
Measure: Median (Standard Deviation); unit: mL
Groups:
- PCI Phase 1: Phase 1 subject undergoing a percutaneous coronary intervention with navigation support of Dynamic Coronary Roadmap
- PCI Phase 2: Not initiated.
Arm/Group | PCI Phase 1 | PCI Phase 2
Number analyzed (Participants) | 23 | 0
mL | 210 (108.77) |

2. Secondary Outcome: Cumulative Dose Area Product (DAP) of Percutaneous Coronary Intervention
Description: No data gathered for the primary outcome. Phase 2 not initiated Only phase 1 data was collected
Time Frame: DAP [mGycm^2] will be determined once, at the end of the Percutaneous Coronary Intervention. There is no patient follow-up.
Population: No data gathered for the primary outcome. Phase 2 not initiated Only phase 1 data was collected
Measure: Median (Standard Deviation); unit: mGy*cm^2
Arm/Group | PCI Phase 1 | PCI Phase 2
Number analyzed (Participants) | 22 | 0
mGy*cm^2 | 116409 (118360) |

3. Secondary Outcome: Cumulative Air-Kerma (AK) of Percutaneous Coronary Intervention
Description: No data gathered for the primary outcome. Phase 2 not initiated Only phase 1 data was collected
Time Frame: AK [mGy] will be determined once, at the end of the Percutaneous Coronary Intervention. There is no patient follow-up.
Population: No data gathered for the primary outcome. Phase 2 not initiated Only phase 1 data was collected
Measure: Median (Standard Deviation); unit: mGy
Arm/Group | PCI Phase 1 | PCI Phase 2
Number analyzed (Participants) | 24 | 0
mGy | 1154 (1022) |

4. Secondary Outcome: Total Fluoroscopy Time of Percutaneous Coronary Intervention
Description: No data gathered for the primary outcome. Phase 2 not initiated Only phase 1 data was collected
Time Frame: Fluoroscopy time [minutes] will be determined once, at the end of the Percutaneous Coronary Intervention. There is no patient follow-up.
Population: No data gathered for the primary outcome. Phase 2 not initiated Only phase 1 data was collected
Measure: Median (Standard Deviation); unit: minutes
Arm/Group | PCI Phase 1 | PCI Phase 2
Number analyzed (Participants) | 24 | 0
minutes | 22 (28.37) |

5. Secondary Outcome: Procedure Efficiency
Description: The endpoint is procedural timing:
  * time from start of procedure (wire introduced into the coronary)
  * end of procedure (start of vascular closure)
  * time until wire placed in distal coronary bed for purpose of intervention
  * time of first stent placement
Time Frame: Patients will be followed from start of interventional procedure (vascular access obtained) until end of the procedure (vascular closure), ranging between 30 minutes and a few hours.
Population: No data gathered for the primary outcome. Phase 2 not initiated Only phase 1 data was collected
Measure: Median (Standard Deviation); unit: minutes
Arm/Group | PCI Phase 1 | PCI Phase 2
Number analyzed (Participants) | 24 | 0
minutes
  The time from start of the procedure until end of the procedure | 46.5 (49.71) |
  The time from start of the procedure until first stent is placed: number analyzed (Participants) | 21 | 0
  The time from start of the procedure until first stent is placed | 24 (19.79) |

6. Other Pre Specified Outcome: Amount of Vessels Treated During Percutaneous Coronary Intervention
Description: Is used as a metric for procedural complexity.
Time Frame: Amount [number] will be determined once, at the end of the Percutaneous Coronary Intervention. There is no patient follow-up.
Population: No data gathered for the primary outcome. Phase 2 not initiated Only phase 1 data was collected
Arm/Group | PCI Phase 2
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Quality of Roadmap Images
Description: The operating physician is asked after the procedure to indicate what the quality and clinical usefulness of those images by scoring on a 5-point rating scale.
Time Frame: Quality [score] will be determined once, at the end of the Percutaneous Coronary Intervention. There is no patient follow-up.
Population: No data gathered for the primary outcome. Phase 2 not initiated Only phase 1 data was collected
Arm/Group | PCI Phase 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Patients were followed-up until discharge through study completion, which was 1 day on average.
Groups:
- PCI Phase 1: Percutaneous coronary interventions with additional imaging provided by the new software package.
  Phase 2 not initiated Only phase 1 data was collected.
Arm/Group | PCI Phase 1
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT02927990/Prot_000.pdf